CLINICAL TRIAL: NCT06187584
Title: Nonopioid Versus Opioid Outpatient Pain Management Following Surgical Fixation of Gartland Type III Supracondylar Humerus Fractures in Children: A Prospective, Randomized Study
Brief Title: SCHF Post-Op Study Between Opioid and Non-Opioid Pain Management
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Caleb Grote, Physician, MD/PhD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000286
Record Dates: First submitted 2023-11-27; First posted 2024-01-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-01

CONDITIONS: Supracondylar Humerus Fracture
MeSH Terms: interventions — oxycodone-acetaminophen; Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Prospective, two-arm, parallel-group, randomized study conducted at a single center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (opioid group) (Active Comparator): Hydrocodone/acetaminophen 0.15mg/kg PO q6 hours PRN with ibuprofen 10mg/kg PO q6 hours PRN
  Interventions: Drug: Hydrocodone/acetaminophen; Drug: Ibuprofen
- Experimental Group (nonopioid group): (Experimental): Acetaminophen 15mg/kg PO q6 hours with ibuprofen 10mg/kg PO q6 hours
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Hydrocodone/acetaminophen — Hydrocodone/acetaminophen 0.15mg/kg PO q6
  Arms: Control Group (opioid group)
Drug: Acetaminophen — 15mg/kg PO q6 hours
  Arms: Experimental Group (nonopioid group):
Drug: Ibuprofen — 10mg/kg PO q6 hours

SUMMARY:
This purpose of this study is to determine the efficacy of nonopioid versus opioid analgesic regimens following surgical fixation of Gartland Type III Supracondylar Humoral Fractures (SCHFs) to assist in the development of a standard outpatient pain management regimen in the treatment of these injuries.

DETAILED DESCRIPTION:
Pain is variably managed in pediatric populations, particularly in the postoperative outpatient setting. The lack of data describing and supporting the safety and efficacy of the use of analgesic drugs in children is a major contributor to this problem. Postoperative prescription opioids have been associated with high rates of morbidity and mortality in children and identified as a pathway to future opioid abuse. With increasing public awareness regarding these issues surrounding opioid use and no evidence to support superior treatment outcomes in children with the use of opioids, there is a pressing need for data to guide healthcare providers in choosing analgesic drugs to treat postoperative pain in pediatric patients.

Prior studies have evaluated the use of nonopioid versus opioid analgesic drugs in the outpatient setting following pediatric ambulatory surgery. These studies found nonopioid analgesics, such as acetaminophen and ibuprofen, to be as equally effective as opioid analgesics, including morphine, codeine and oxycodone. Further, the use of nonopioid analgesics was associated with significantly fewer side effects. These findings imply that nonopioid analgesics may be a superior initial therapy following ambulatory surgery.

However, no study has evaluated the use of nonopioid versus opioid analgesic regimens in the outpatient setting following surgical fixation of supracondylar humerus fractures (SCHFS). SCHFs are the second most common fracture in children, often requiring urgent surgical intervention. Despite their frequency, there is no standard for postoperative outpatient pain management in the treatment of these injuries.

Almost all SCHFs can be described according to the Gartland classification. The Gartland classification delineates three types of SCHFs. Gartland type I fractures are nondisplaced and do not require surgical intervention, while Gartland type II fractures are angulated, but maintain an intact posterior cortex. These may or may not require surgical intervention. However, Gartland type III fractures are completely displaced with no posterior cortical contact and require surgical intervention with either closed reduction and percutaneous pinning (CRPP) or open reduction with percutaneous pinning (ORPP). This study will look at only Gartland type III SCHFs because they necessitate surgical intervention, most commonly CRPP.

Investigators hypothesize that there is no difference in daily pain levels for nonopioid analgesic regimens compared to opioid analgesic regimens in management of post-operative pain in the outpatient period following surgical fixation of Gartland type III supracondylar humerus fracture in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Children's Mercy Hospital
* Patients 48-119 months of age
* Closed and completely displaced Gartland type III SCHFs (ICD-10 codes: S42.411A, S42.412A and S42.413A)

Exclusion Criteria:

* Patients younger than 48 months of age or older than 120 months of age
* Nondisplaced SCHFs (ICD-10): S42.414-, S42.415- and S42.416-)
* Open and completely displaced Gartland type III SCHFs (ICD-10: S42.411B, S42.412B and S42.413B)
* Injury requiring open reduction and/or vascular injury requiring treatment
* Patients presenting with additional injuries
* Patients with known allergy to medications used in this study
* Patients receiving regular treatment with opioids or NSAIDs
* Patients with underlying medical issues affecting cognitive status
* Patients with hepatic, gastrointestinal, renal or hematologic disease/disorders
* Children that are wards of the state, prisoners or of CM employees
* Non-English speaking families
* Patients not admitted before and after surgery
* Fractures not surgically treated within 18 hours of injury
* Use of local anesthetic at surgical site

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be subject reported pain level using the Wong-Baker Faces Pain Scale. | At the relative same time each day on postoperative days 1-5 (i.e., five follow-up measures).
  The subject reported pain level using the scale 0-10, will be measured at the time of discharge (i.e., baseline measure).

SECONDARY OUTCOMES:
Parent satisfaction with (subject) child's pain control | Two hours post intervention and everyday at the same time as the initial response for five consecutive days post intervention
  Using the Likert scale, "very dissatisfied, dissatisfied, neutral, satisfied, very satisfied" options, the investigators ask families to rate the satisfaction of their child's pain control daily for 5 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital & Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] Alkhoury F, Knight C, Stylianos S, Zerpa J, Pasaron R, Mora J, Aserlind A, Malvezzi L, Burnweit C. Prospective Comparison of Nonnarcotic versus Narcotic Outpatient Oral Analgesic Use after Laparoscopic Appendectomy and Early Discharge. Minim Invasive Surg. 2014;2014:509632. doi: 10.1155/2014/509632. Epub 2014 Apr 14. PMID 24834350
- [Background] Tubbs RS, Law C, Davis D, Shoja MM, Acakpo-Satchivi L, Wellons JC 3rd, Blount JP, Oakes WJ. Scheduled oral analgesics and the need for opiates in children following partial dorsal rhizotomy. J Neurosurg. 2007 Jun;106(6 Suppl):439-40. doi: 10.3171/ped.2007.106.6.439. PMID 17566399
- [Background] Tobias JD. Acute pain management in infants and children-Part 1: Pain pathways, pain assessment, and outpatient pain management. Pediatr Ann. 2014 Jul;43(7):e163-8. doi: 10.3928/00904481-20140619-10. PMID 24977679
- [Background] Tobias JD. Acute pain management in infants and children-Part 2: Intravenous opioids, intravenous nonsteroidal anti-inflammatory drugs, and managing adverse effects. Pediatr Ann. 2014 Jul;43(7):e169-75. doi: 10.3928/00904481-20140619-11. PMID 24977680
- [Background] Poonai N, Datoo N, Ali S, Cashin M, Drendel AL, Zhu R, Lepore N, Greff M, Rieder M, Bartley D. Oral morphine versus ibuprofen administered at home for postoperative orthopedic pain in children: a randomized controlled trial. CMAJ. 2017 Oct 10;189(40):E1252-E1258. doi: 10.1503/cmaj.170017. PMID 29018084
- [Background] Dorkham MC, Chalkiadis GA, von Ungern Sternberg BS, Davidson AJ. Effective postoperative pain management in children after ambulatory surgery, with a focus on tonsillectomy: barriers and possible solutions. Paediatr Anaesth. 2014 Mar;24(3):239-48. doi: 10.1111/pan.12327. Epub 2013 Dec 11. PMID 24330523
- [Background] Austin AE, Shanahan ME, Zvara BJ. Association of childhood abuse and prescription opioid use in early adulthood. Addict Behav. 2018 Jan;76:265-269. doi: 10.1016/j.addbeh.2017.08.033. Epub 2017 Sep 1. PMID 28869906
- [Background] Dart RC, Surratt HL, Cicero TJ, Parrino MW, Severtson SG, Bucher-Bartelson B, Green JL. Trends in opioid analgesic abuse and mortality in the United States. N Engl J Med. 2015 Jan 15;372(3):241-8. doi: 10.1056/NEJMsa1406143. PMID 25587948
- [Background] Cartabuke RS, Tobias JD, Taghon T, Rice J. Current practices regarding codeine administration among pediatricians and pediatric subspecialists. Clin Pediatr (Phila). 2014 Jan;53(1):26-30. doi: 10.1177/0009922813498151. Epub 2013 Aug 5. PMID 23922249
- [Background] Marquis, C.P., Cheung, G., Dwyer, J.S.M., et al. "Supracondylar fractures of the humerus". Current Orthopaedics. 2008;22:62-69.
- [Background] Chaturvedi H, Khanna V, Bhargava R, Vaishya R. Predictive factors determining outcomes in pulseless limb in paediatric supracondylar fractures of humerus. J Clin Orthop Trauma. 2018 Mar;9(Suppl 1):S92-S96. doi: 10.1016/j.jcot.2017.10.009. Epub 2017 Oct 31. PMID 29628707
- [Background] Woon, C., Souder, C. and Skaggs, D. "Supracondylar Fracture - Pediatric". Orthobullets. https://www.orthobullets.com/pediatrics/4007/supracondylar-fracture--pediatric. (17 July 2018).
- [Background] Flynn JC, Matthews JG, Benoit RL. Blind pinning of displaced supracondylar fractures of the humerus in children. Sixteen years' experience with long-term follow-up. J Bone Joint Surg Am. 1974 Mar;56(2):263-72. No abstract available. PMID 4375679
- [Background] The Wong-Baker FACES Foundation: Faces of Pain Care. c2016. Published 2018. Wong-Baker FACES Foundation. [Accessed 11 Oct. 2018]. http://wongbakerfaces.org.